CLINICAL TRIAL: NCT07006025
Title: Phase 1 Study of Oral Tetrahydrouridine-Decitabine to Treat Relapsed or Refractory Myelodysplastic Syndromes
Brief Title: A Study of Oral Tetrahydrouridine-Decitabine in Relapsed or Refractory Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Treebough Therapies (Industry)
Collaborators: EpiDestiny, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00001
Record Dates: First submitted 2025-05-20; First posted 2025-06-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: MDS
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: Single arm, open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): Oral capsules of THU followed 1 hour later by decitabine
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Oral tetrahydrouridine and oral decitabine capsule
  Other Names: Decagen

SUMMARY:
The goal of this clinical trial is to learn about the safety and effectiveness of the combination drug Tetrahydrouridine (THU) and decitabine (DEC) to treat patients with relapsed or refractory myelodysplastic syndrome. The main questions it aims to answer are:

* Does the combination drug exhibit hematological and nonhematological toxicity?
* Does the combination drug improve health status and reduce the number of days of hospitalization?

Participants will:

* Take tetrahydrouridine and decitabine once a week for 24 weeks
* Visit the clinic once every 4 weeks for checkups and tests
* Keep a diary of their symptoms

DETAILED DESCRIPTION:
This is a single-arm, open-label Phase 1 study of oral THU/decitabine to treat relapsed or refractory MDS. Patients will be treated for 24 weeks in the absence of clear evidence of progressive disease. The primary endpoint is safety. The secondary endpoints will include assessment of response rates by International Working Group (IWG) criteria, quality of life (QoL), and number of days of hospitalization. DNA-methyltransferase 1 (DNMT1) protein levels will be measured in bone marrow and peripheral blood white cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of MDS that has received one or more prior standard therapies and is relapsed or refractory
* Patients must be 18 years of age or older
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3
* Patients must have adequate end-organ function
* Patient's body weight must be ≥ 41 kg
* Subjects must be able to understand and willing to sign a written informed consent document and complete study-related procedures.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL)
* Prior treatment with ≥4 28-day cycles of parenteral or oral decitabine
* No other disease-directed therapy, save for hydroxyurea, including experimental or investigational drug therapy for 14 days prior to study entry (hydroxyurea should be discontinued ≥24 hours prior to initiation of study drug)
* Requiring concomitant treatment with drugs that are cytidine deaminase (CDA) substrates and/or inhibitors, e.g., cytarabine, 5-azacytidine, gemcitabine
* Currently pregnant or breastfeeding. Females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment start.
* Uncontrolled intercurrent illness that could limit life expectancy or ability to complete study correlates
* Women of Childbearing Potential (WOCBP) who are unwilling to agree to use dual contraceptive measures (i.e., hormonal or barrier method of birth control; abstinence, condom) prior to study entry, for the duration of study participation, and until 6 months after taking the last dose of THU/decitabine
* Sexually active male who is unwilling to use a condom when engaging in any sexual contact with a WOCBP, beginning at the screening visit and continuing until 6 months after taking the last dose of THU/decitabine
* 9. Patients with uncontrolled active human retrovirus (HIV) infection, as this will further increase the risk for opportunistic infections. However, patients with HIV with undetectable viral load by polymerase chain reaction (PCR), without opportunistic infection, and on a stable regimen of antiretroviral therapy are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
White blood cell measurement | every 4 weeks
  Measure neutrophils count
Platelet count | every 4 week
  Measure platelets in the blood

SECONDARY OUTCOMES:
Response for high-risk MDS | every 4 weeks
  Measure using International Working Group (IWG) 2023 response criteria
Hospitalization | every 4 weeks
  Record the number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Goldfinger, MD, Principal Investigator — Montefiore/Einstein Cancer Center
Locations (1):
- Montefiore Einstein Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No